CLINICAL TRIAL: NCT03069898
Title: Evaluation of the TRUE Dads Intervention
Brief Title: TRUE Dads: Evaluation of an Intervention Focusing on Father Involvement, Co-parenting, and Employment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: It's My Community Initiative (Other)
Responsible Party: Principal Investigator, Philip A. Cowan, Professor of Psychology Emeritus, University of California, Berkeley, It's My Community Initiative
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2016-08-9047
Record Dates: First submitted 2017-02-28; First posted 2017-03-03 (Actual); Last update posted 2020-08-26 (Actual); Status verified 2020-08

CONDITIONS: Father-Child Relations
Keywords: Marital relationship

STUDY DESIGN:
Intervention Model Description: Paraticipants are randomly assigned to intervention (TRUE Dads) and Control tracks, assessed at Baseline and again one year later. The intervention primarily involves attendance at 12 3-hour workshops for fathers and their co-parents.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TRUE Dads program track (Experimental): In the TRUE Dads program, fathers and co-parents begin with a Core workshop meeting weekly for 6 weeks. After a check-in, a male-female group leader team focuses on a single topic that represents one of the three main goals of the project as a whole: Co-parenting relationships, Parenting, or Employment and financial stability. From 10 to 18 couples, seated at small tables in a large room, hear mini-lectures, watch videos, and engage in interactive exercises. Fathers then choose to attend one of three intensive workshops focused on couple relationships OR parenting OR economic self-sufficiency meeting 3 hours per week for the next 6 weeks. On an as-needed basis, fathers may be referred for employment programs and fathers and co-parents may be referred for mental health or other services.
  Interventions: Behavioral: TRUE Dads
- Control condition study track (No Intervention): Participants (fathers and co-parents) complete intake interview and fill out Baseline survey. They fill out follow-up survey one year later

INTERVENTIONS:
Behavioral: TRUE Dads — The TRUE Dads intervention consists of a set of 12 3-hour workshops that focus on enhancing fathers' role as co-parent, parent, and provider
  Arms: TRUE Dads program track

SUMMARY:
With an emphasis on 12 3-hour group workshops, the TRUE Dads fatherhood intervention program focuses on establishing or strengthening three of men's key roles in the family: 1) their role as providers, through fostering employment and economic self-sufficiency, 2) their role as fathers, in building and maintaining positive engagement with their children, and 3) their role in having and keeping a positive relationship with their co-parenting partner (wife, intimate partner, or other co-parent). The study is a randomized clinical trial that compares participants in a program track with participants a study track (no treatment control group) over a one-year period.

DETAILED DESCRIPTION:
Interventions to strengthen men's roles as providers, as fathers, and as co-parents have typically been addressed in separate intervention and research silos. The TRUE Dads program proposes a unique integration of employment, fathering, and co-parenting services, with the overarching goal of strengthening fathers and the family unit by: 1) increasing fathers' economic stability and self-sufficiency, 2) enhancing the quantity and quality of father's engagement with their children, 3) improving the quality of the collaborative relationship between fathers and mothers or men and their co-parenting partners, 4) improving the relationship quality of fathers in their intimate partner relationships (with the co-parent or new partner), and 5) positively affecting children's behavior and development.

Twelve hundred fathers will be recruited for the study. After an initial interview of the fathers and their co-parenting partners, who will complete Baseline survey, 720 of the 1,200 fathers and co-parents will be assigned to the TRUE Dads intervention (Program track), and 480 to a no-treatment control condition (Study track). Participants will be informed that the program consists of participation in a series of 12 three-hour meetings. Those 12 sessions include six meetings covering a core fatherhood curriculum, attended with the co-parent, combined with one of three intensives selected by the father: a) six sessions with an emphasis on employment, b) six sessions with an emphasis on building healthy romantic relationships with the co-parent, or c) six sessions with an emphasis on parenting with a participating co-parent. Participants in the Program track may be referred for additional employment, mental health, or other needed services. Both program and control participants (fathers and co-parents) will fill out a Follow-up survey one year from their entrances into the study.

ELIGIBILITY:
Inclusion criteria:

This study begins with a focus on fathers. We are initially recruiting men who:

* Are 18 or older
* Are residing in Oklahoma County/Metro
* Are expecting a child or already have a child age (0-12), with an emphasis on 0-6,
* Have spent time with the child the prior month (or with mother if expecting)
* Are English-speaking. Have not previously participated in the Family Expectations program offered by Public Strategies (Oklahoma) in the last 3 years

Exclusion criteria:

Because this an intervention for fathers that attempts to improve the relationship with the fathers' co-parent, we are accepting fathers only if the co-parent agrees to attend at least the first 6 workshops. In pilot trials, almost all the co-parents are women (wives, intimate partners, grandmothers), but a few are men (the fathers' father, brother, intimate partner)

-

Exclusion Criteria:

* Either or both partners have taken part in the Family Expectations project during the past three years, located in the same building, run by Public Strategies

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — The primary focus of the study is on fatherhood, so the entrance to the study begins with fathers. But each father must bring the primary person with whom he is co-parenting his child -- wife, romantic partner, friend, mother. Usually the co-parent is a woman, but occasionally a man (father's father, intimate partner).
Enrollment: 2084 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Father/Co-parent relationship quality | Change or maintenance of positive behavior relative to the control group will be assessed at Baseline and 1 year post Baseline.
  This outcome will be measured by a composite of self-report survey items filled out by fathers and co-parents, assessing perceptions of co-parent relationship quality, communication and conflict management abilities. High scores indicate relationship distress.
Father involvement | Change or maintenance of positive behavior relative to the control group will be assessed at Baseline and 1 year post Baseline.
  This outcome will be measured by a composite of self-report survey items filled out by both fathers and co-parents, assessing fathers' involvement in childcare tasks, time spent in specific activities with target child, parenting styles, and parenting behaviors. High scores indicate positive father involvement
Child well-being | Change or maintenance of positive behavior relative to the control group will be assessed at Baseline and 1 year post Baseline.
  This outcome will be measured by a composite of self-report survey items filled out by fathers and co-parents, assessing child temperament, externalizing behavior problems (aggression, hyperactivity) and internalizing behavior problems (anxiety, depression, shy/withdrawn behavior). High scores indicate more behavior problems.
Economic Self-sufficiency | Change or maintenance of positive behavior relative to the control group will be assessed at Baseline and 1 year post Baseline.
  This outcome will be measured by a composite of self-report survey items filled out by fathers and co-parents, assessing employment status, income, behaviors to find a job or acquire new job skills. High scores indicate more positive economic achievements and more positive attitudes
Parents adjustment and distress | change or maintenance of positive behavior relative to the control group will be assessed at Baseline and 1 year post Baseline.
  This outcome will be measured by a composite of self-report measures of symptoms of depression (Center for Epidemiological Studies in Depression, CES-D) and anxiety (from the Brief Symptom Inventory). High scores indicate personal distress.

CONTACTS AND LOCATIONS:
Overall Officials: Philip A. Cowan, PhD, Principal Investigator — It's My Community Initiative
Locations (1):
- It's My Community Initiative, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Cowan PA, Cowan CP, Gillette PF. TRUE Dads: The impact of a couples-based fatherhood intervention on family relationships, child outcomes, and economic self-sufficiency. Fam Process. 2022 Sep;61(3):1021-1044. doi: 10.1111/famp.12748. Epub 2022 Jan 10. PMID 35014030